CLINICAL TRIAL: NCT06659978
Title: Missing Touch 1: Human Factors Validation and Acceptability Testing of a Neuro-engineered C-tactile Stimulation Device
Brief Title: Human Factors Validation and Acceptability Testing of a Stimulation Device
Acronym: NICU-TAC
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool John Moores University (Other); Liverpool Women's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UoL001661
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Human Factors; Acceptability; Tolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infants: Well, infants born between 34 and 42 weeks.
  Interventions: Device: Device tolerance; Other: Acceptability questionnaire

INTERVENTIONS:
Device: Device tolerance — After being fed (breastmilk or formula), video will be turned on and the infant is placed on the Gentle Touch Stimulator (GTS) in deactivated mode. After a baseline period of 5- minutes the device will be activated. It will be deactivated after 10 minutes or earlier if there are any signs of distress from the infant. A 10-minute washout observation period will be followed.
  Higher levels of comfort will be considered as fewer instances of stress behaviours. The sessions will be videoed, and coded at a later date using Observation of infant behaviours.
Other: Acceptability questionnaire — Parental and clinical staff acceptability of the device assessed by interviewing person(s) of parental responsibility and clinicians involved in the trial. Interviews will be conducted by researcher following the intervention.

SUMMARY:
Our team have developed a mattress topper, consisting of rubber tubes attached side to side that are deflated and inflated, mimicking dynamic touch and optimal CT stimulation (3cm/s). It is connected to a microprocessor control unit and a vacuum supply. By controlling the interval between the vacuum applied to each tube in the device it generates a flow sequence as each tube relaxes back to its original state. This will feel like a stroking across the skin - but non-frictional, thereby minimising the risk of friction related skin damage.

The device is placed on top of a standard mattress in a neonatal cot. It has been manufactured in line with European Union (EU) safety requirements. It has been calibrated to mimic optimal CT fibre activation at 3cm/s, in line with previous touch intervention studies (Gursul et al., 2018; Manzotti et al., 2019). The device is made from silicone and is fully waterproof. A cleaning protocol will be implemented between each use for infection control. The waterproof sheet will be covered by a standard cot sheet.

DETAILED DESCRIPTION:
New-born infants are subject to several novel experiences that cause physiological, biochemical and behavioural indicators of stress; even routine and common events such as handling, changing a diaper or being bathed can induce a stress response. Tactile interventions such as skin-to-skin touch and 'still containment hold' are widely used in clinical care with apparent positive results, such as lower mean respiratory heart rate and pain measures, and higher oxygen saturation (Boundy et al., 2016; Pineda et al., 2017); yet, dynamic touch interventions have reported to be more beneficial than static touch interventions (Field, Diego, Hernandez-Reif, Deeds, & Figuereido, 2006; Manzotti et al., 2019; Vickers, Ohlsson, Lacy, & Horsley, 2004).

A distinct class of unmyelinated C-fibre sensory neurons called C-tactile afferents (CT), found exclusively in the hairy skin of the body, that respond optimally to gentle stroking touch at a velocity of ~3cm/s, are hypothesised to process the pleasant and social rewarding properties of touch (Olausson et al., 2010, McGlone et al., 2014). CT fibre activation also plays a role in pain inhibition (Gursul et al., 2018; Habig et al., 2017; Liljencrantz et al., 2017) and may also be linked to the development of self-regulation (Van Puyvelde, Gorissen, Pattyn, & McGlone, 2019), thereby serving a neuroprotective function for the developing infant brain.

Touch induced-analgesia such as skin-to-skin contact and breastfeeding are also considered as standard care non-pharmacological interventions for procedural pain in infants (Campbell-Yeo et al., 2019; Chang, Filoteo, & Nasr, 2020). However, dynamic touch is not currently acknowledged as a non-pharmacological intervention in the UK.

Touch is the first sense to develop in utero at approximately 8-weeks gestational age and is the most mature sense postnatally (Marx & Nagy, 2015). The benefits of touch are now widely recognised in postnatal care with the World Health Organization (2019) recommending that term infants engage in skin-to-skin contact with their mother or carer for at least an hour after birth due to the physiological benefits for both infant and mother.

There is limited research into the underlying mechanism behind the physiological benefits of touch, either in-utero or post-partum; however, it is hypothesised that foetal movements cause the amniotic fluid to elicit movement of lanugo (fine hair), which activates specific nerve fibres - C-Tactile afferents (CTs) to facilitate growth regulation (Bystrova, 2009).

CTs signal the affective component of touch (Löken, Wessberg, Morrison, McGlone, & Olausson, 2009; McGlone, Cerritelli, Walker, & Esteves, 2017). Found exclusively in hairy skin they project to the insular cortex (Olausson et al., 2002), part of the brain's self-regulation system and associated with emotional processing (Dalgleish, 2004). Microneurography, a method employed to visualise and record the traffic of nerve impulses, from CTs find that they respond optimally to low force and velocity dynamic touch delivered at ~ 3cm/sec at skin temperature (Löken et al., 2009), supporting the hypothesis of the social function for the nerve in nurture, grooming and affiliative behaviours.

A recent study carried out with preterm infants in a Neonatal Intensive Care Unit (NICU) found that dynamic touch, delivered at CT optimal speed, reduced heart rate and increased blood oxygenation levels in neonates (Manzotti et al., 2019). Should the hypothesis be accepted in this study it will offer insight into some of the mechanisms behind the physiological advantages of touch, leading to the improvement of neurodevelopmental outcomes for newborns e.g., during painful procedures. However, there are instances where infants are deprived of touch, such as lack of skin integrity and risk of infections, lack of parental presence and disorders such as foetal alcohol syndrome or neonatal abstinence syndrome. This series of studies is aimed at individuals who are deprived of touch - it is not seen as a replacement for maternal/carer touch.

Here we will investigate the tolerability of the device-delivered tactile stimulation at CT-optimal velocity by measuring physiological indicators of stress in infants, as determined by heart rate and blood oxygenation, and assessment of stress behaviours.

ELIGIBILITY:
Inclusion Criteria:

* Infant is born between 34- and 42-weeks gestational age.
* Infant an in-patient at LWH based on the low dependency unit or post-natal ward.
* Infant is born from a low-risk pregnancy with no concerns identified antenatally or postnatally.
* Infant has been identified as eligible by neonatal clinician (junior doctor or advanced neonatal nurse practitioner).
* Written consent has been obtained from the person(s) with parental responsibility.
* Infant has been normoglycaemic since birth or for at least 24 hours.

Exclusion Criteria:

* Known genetic condition or undergoing investigation for a suspected genetic condition.
* Previously admitted to high dependency or intensive care.
* Has received invasive respiratory support.
* Has received any treatment for seizures.
* Is receiving phototherapy.
* Is receiving caffeine.
* Concerns about feeding (e.g., a condition that may interfere with feeding such as cleft palate or any tube feeding at the time of the study) NB tongue tie is NOT an exclusion criterion.
* Needing any support for thermoregulation (in incubator or using "hot cot")
* Clinical instability in the judgment of nurses/midwives and paediatricians looking after the baby and mother.

Ages: 34 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Well infant born between 34 and 42 weeks in the low dependency unit or postnatal ward.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Infant device tolerance | 25 minutes
  Infant's physiological responses to the device are measured by heart rate and blood oxygenation

SECONDARY OUTCOMES:
Infant comfort levels | 25 minutes
  Higher levels of comfort will be considered as fewer instances of stress behaviours. The sessions will be videoed, and coded at a later date using Observation of infant behaviours.
Parental and clinical staff acceptability | 15 minutes
  Assessed by interviewing person(s) of parental responsibility and clinicians involved in the trial

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Liverpool John Moores University, Liverpool
  - Liverpool Womens Hospital Trust, Liverpool
  - University of Liverpool, Liverpool

IPD SHARING:
Plan to Share IPD: No